CLINICAL TRIAL: NCT01406847
Title: Central Mechanisms of Body Based Intervention for Musculoskeletal Low Back Pain
Brief Title: Central Mechanisms of Intervention for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201602462-N; 1R01AT006334-01 (NIH); 439-2010 (Other: UF legacy)
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Low Back Pain
Keywords: Spinal Manipulation; Body-based intervention; Experimental pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spinal Manipulation (Experimental): High-velocity manual technique applied to the pelvis with the participant in supine
  Interventions: Other: Spinal Manipulation
- Static Touch (Sham Comparator): Practitioner hands are placed on the lumbar spine with the participant in prone.
  Interventions: Other: Static Touch
- Spinal Mobilization (Active Comparator): Oscillation of the third lumbar level performed with the participant in prone
  Interventions: Other: Spinal Mobilization

INTERVENTIONS:
Other: Spinal Manipulation — High velocity low amplitude joint-biased intervention
  Other Names: SMT
  Arms: Spinal Manipulation
Other: Spinal Mobilization — Low velocity, large amplitude oscillating joint biased technique
  Other Names: Mobilization; Mobs
  Arms: Spinal Mobilization
Other: Static Touch — The investigators maintains hand contact with both hands over the lumbar area of the participant
  Arms: Static Touch

SUMMARY:
Body-based interventions have consistently shown clinical effectiveness in patients with back pain. The primary objective for this study is to compare the effect of body-based interventions commonly used in the management of low back pain on behavioral and cortical measures of pain sensitivity and central sensitization of pain. Participants will be randomly assigned to receive one of the interventions or be in a control group. The central hypothesis for this proposal is that spinal manipulation, a specific form of body-based intervention, inhibits central sensitization of pain normalizing pain sensitivity more rapidly than other interventions. The completion of the proposed study will elucidate underpinning mechanisms of body-based interventions. Identification of these mechanisms will improve the clinical application and utilization of these interventions in the management of musculoskeletal pain conditions, especially back pain.

DETAILED DESCRIPTION:
170 participants will be randomly assigned to receive one of the interventions or be in a control group. The investigators will use of a model of experimentally induced low back pain to investigate the effects of manipulative and body-based interventions in acute onset low back pain without some of the clinical confounds. The investigators will collect fMRI and psychophysical data about pain sensitivity before and after the induction of pain, and before and after interventions for that pain.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 40 years
* able to read and understand spoken English

Exclusion Criteria:

* Previous participation in a conditioning program specific to trunk extensors in the past 6 months
* Any report of back or leg pain in the past 3 months
* Any chronic medical conditions that may affect pain perception (e.g., diabetes, high blood pressure, fibromyalgia, headaches), kidney dysfunction, muscle damage, or major psychiatric disorder
* History of previous injury including surgery to the lumbar spine, renal malfunction, cardiac condition, high blood pressure, osteoporosis, or liver dysfunction
* Consumption of any drugs (e.g., caffeine, alcohol, theophyline, tranquilizers, antidepressants) that may affect pain perception or hydration status from 24 hr. before participation until completion of the investigation
* Performance of any intervention for symptoms induced by exercise and before the termination of their participation or the protocol
* Recent illness
* Any contraindication to MRI e.g.: pacemakers, metal implants which are not MRI compatible (e.g. aneurysm clip), pregnancy and severe claustrophobia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2012-08; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Immediate change in temporal sensory summation | 10 minutes post-intervention
  We will use both behavioral (ratings) and cortical (using fMRI) measures of temporal sensory summation.
Change in temporal sensory summation | 48 hours post-intervention
  The change temporal sensory summation (determined using quantitative sensory testing and fMRI) will be calculated from pre-intervention to 48 hours post-intervention

SECONDARY OUTCOMES:
Change in Physical Impairment Index | 48 hours post-intervention
  Physical Impairment Index is a group of tests including trunk and limb range of motion, muscle tenderness and abdominal muscle performance

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Bishop, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States